CLINICAL TRIAL: NCT05003713
Title: A Phase I Adaptive Dose, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally Administered CORT125236 in Healthy Subjects, With an Optional Pharmacological Effects Cohort
Brief Title: Single and Multiple Ascending Dose Study of CORT125236 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: CORT125236-150; 2021-001407-32 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1: SAD Cohorts A through F CORT125236 (Experimental): Cohorts will receive a single dose of CORT125236 lipid capsule formulation by mouth on Day 1 in a fasted or fed state. Cohort A will receive a 20-mg dose in a fasted state. Cohort B will receive a ≤3-fold increase in dose from Cohort A in a fasted state; the dose level and dose regimen (whether to split the dose) will be determined after evaluation of safety and PK data for Cohort A. Subsequent cohorts will receive a ≤3-fold increase in CORT125236 dose from the previous cohort in a fasted or fed state; the dose level, dose regimen, and prandial state will be determined after evaluation of safety and PK data from previous cohorts.
  Interventions: Drug: CORT125236
- Part 1: SAD Cohorts A through F Placebo (Placebo Comparator): Cohorts will receive a single dose of placebo matching CORT125236 lipid capsule formulation by mouth on Day 1. The dose regimen and prandial state will be the same as those for the cohort members receiving CORT125236.
  Interventions: Drug: Placebo matching CORT125236
- Part 2: MAD Cohorts A through D CORT125236 (Experimental): Cohorts will receive once- or twice-daily doses of CORT125236 lipid capsule formulation by mouth for 14 days. The anticipated exposure will not exceed the highest exposure considered safe and well-tolerated during Part 1. The dose level, dose schedule, and prandial state for each cohort will be determined after evaluation of safety and PK data from Part 1 and preceding Part 2 cohorts.
  Interventions: Drug: CORT125236
- Part 2: MAD Cohorts A through D Placebo (Placebo Comparator): Cohorts will receive once- or twice-daily doses of placebo matching CORT125236 lipid capsule formulation by mouth for 14 days. The dose regimen and prandial state will be the same as those for the cohort members receiving CORT125236.
  Interventions: Drug: Placebo matching CORT125236
- Part 3: Single Dose Pharmacodynamic Effect (Experimental): In Period 1, participants will receive a single dose of prednisone 25 mg (20 mg + 5 mg) tablet by mouth on Day 1 in a fasted or fed state. After a 7-day washout, in Period 2, participants will receive a single dose of prednisone as in Period 1 plus a single dose of CORT125236 lipid capsule formulation by mouth on Day 1 in a fasted or fed state. The dose of CORT125236 and the prandial state will be determined after evaluation of safety and PK data from Part 1. Part 3 of the study is optional.
  Interventions: Drug: CORT125236; Drug: Prednisone

INTERVENTIONS:
Drug: CORT125236 — CORT125236 Lipid Capsule Formulation 10-60 mg for oral administration
  Arms: Part 1: SAD Cohorts A through F CORT125236; Part 2: MAD Cohorts A through D CORT125236; Part 3: Single Dose Pharmacodynamic Effect
Drug: Placebo matching CORT125236 — Placebo matching CORT125236 Lipid Capsule Formulation 10-60 mg for oral administration
  Arms: Part 1: SAD Cohorts A through F Placebo; Part 2: MAD Cohorts A through D Placebo
Drug: Prednisone — Prednisone tablet 25 mg (20 mg + 5 mg tablets) for oral administration
  Arms: Part 3: Single Dose Pharmacodynamic Effect

SUMMARY:
This is a 3-part, first-in-human study of single ascending doses (SAD; Part 1) and multiple ascending doses (MAD; Part 2) of CORT125236 in healthy participants; Part 3 is optional, to investigate whether CORT125236 ameliorates the effects of prednisone on various pharmacodynamic (PD) endpoints. The 3 parts may not be conducted entirely sequentially provided that this is justified by the pharmacokinetic (PK) and safety data obtained from completed cohorts. The first MAD cohort will not start until data are available from at least 3 SAD levels to allow MAD administration to proceed. The decision on whether to start Part 3 can be made at any point after completion of 3 SAD levels, and will be based on achieving sufficiently high plasma CORT125236 exposure in Part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0 to 30.0 kg/m^2, inclusive
* Body weight ≤102 kg
* Willing to consume a high-fat breakfast, including pork
* Adheres to the contraception requirements of the protocol
* Additional criteria apply.

Exclusion Criteria:

* Received any investigational drug or device in a clinical research study within 90 days
* Evidence of current severe acute respiratory syndrome (SARS-CoV-2) infection
* History of any drug or alcohol abuse in the past 2 years; a confirmed positive drugs of abuse test result
* Regular alcohol consumption; a confirmed positive alcohol breath test at screening
* Current smoker; a confirmed positive breath carbon monoxide reading; current user of e-cigarettes and nicotine replacement products in the last 6 months
* Female of childbearing potential, pregnant, or breastfeeding
* Male participant with pregnant or lactating partners
* Clinically significant abnormal clinical chemistry, hematology or urinalysis result
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV)
* Active renal and/or hepatic disease
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, respiratory, gastrointestinal (GI), neurological or psychiatric disorder
* Any form of cancer in the 5 years (exceptions apply)
* History of adrenal insufficiency
* Have a condition that could be aggravated by glucocorticoid antagonism
* Donation or loss of greater than 400 mL of blood or plasma within the previous 3 months
* Currently using glucocorticoids or have a history of systemic glucocorticoid use in the last 12 months or 3 months for inhaled products
* Additional criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events | Part 1 SAD Cohorts: up to Day 12; Part 2 MAD Cohorts: up to Day 25; Part 3 Cohort: up to Day 19

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CORT125236 | Before dosing and at pre-specified time points up to Day 5 (Part 1 SAD Cohorts), or up to Day 18 (Part 2 MAD Cohorts)
Time of Cmax (Tmax) of Plasma CORT125236 | Before dosing and at pre-specified time points up to Day 5 (Part 1 SAD Cohorts), or up to Day 18 (Part 2 MAD Cohorts)
Apparent Elimination Half-life (t1/2) of Plasma CORT125236 | Before dosing and at pre-specified time points up to Day 5 (Part 1 SAD Cohorts), or up to Day 18 (Part 2 MAD Cohorts)
Area Under the Plasma Concentration-time Curve (AUC) of CORT125236 | Before dosing and at pre-specified time points up to Day 5 (Part 1 SAD Cohorts), or up to Day 18 (Part 2 MAD Cohorts)
Serum Cortisol Concentration | Before dosing on Days 1 and 14 (Part 2 MAD Cohorts)
Plasma Adrenocorticotropic Hormone (ACTH) Concentration | Before dosing on Days 1 and 14 (Part 2 MAD Cohorts)
Eosinophil Count | Before dosing and at pre-specified time points up to 24 hours after dosing (Part 3, Periods 1 and 2 PD Cohort)
Lymphocyte Count | Before dosing and at pre-specified time points up to 24 hours after dosing (Part 3, Period 1 and 2 PD Cohort)
Neutrophil Count | Before dosing and at pre-specified time points up to 24 hours after dosing (Part 3, Period 1 and 2 PD Cohort)
Serum Osteocalcin Concentration | Before dosing and at pre-specified time points up to 24 hours after dosing (Part 3, Period 1 and 2 PD Cohort)
Plasma Glucose | 4 hours after dosing and immediately prior to a high-carbohydrate lunch, and approximately 2 hours after starting the lunch (Part 3, Period 1 and 2 PD Cohort)
Serum Insulin | 4 hours after dosing and immediately prior to a high-carbohydrate lunch, and approximately 2 hours after starting the lunch (Part 3, Period 1 and 2 PD Cohort)
Plasma Tumor Necrosis Factor Alpha (TNF-α) Concentration following ex vivo Lipopolysaccharide (LPS) Stimulation | Before dosing and 1, 2, and 4 hours after dosing (Part 3, Periods 1 and 2 PD Cohort)
Plasma Interleukin-1 Beta (IL-1β) Concentration following ex vivo LPS Stimulation | Before dosing and 1, 2, and 4 hours after dosing (Part 3, Periods 1 and 2 PD Cohort)

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Hunt, Ph.D., Study Director — Corcept Therapeutics
Locations (1):
- Site 01, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No